CLINICAL TRIAL: NCT05887947
Title: Impact of E-cigarette Nicotine Concentration on Compensation, Cigarette Smoking, and Biomarkers of Exposure and Harm in Diverse Smokers
Brief Title: Impact of E-cigarette Nicotine Concentration on Compensation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 147694; K01DA054995 (NIH)
Record Dates: First submitted 2023-05-12; First posted 2023-06-05 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: We will conduct a 2x2 crossover study and utilize linear mixed effects models to assess differences in total inhaled volume between 1.8% and 5% nicotine concentration. Phase 1 (P1): 2-visit human laboratory trial with double-blind, randomized crossover design. Phase 2 (P2): 6-week, randomized substitution trial. Participants in P2 will be the same participants that completed P1.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Phase 1 (P1): 2-visit human laboratory trial with double-blind, randomized crossover design. Phase 2 (P2): 6-week, randomized open-label substitution trial. No blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 5% Nicotine E-cigarette Followed by 1.8% Nicotine E-cigarette (Experimental): At lab visit 1 participants receive 5% electronic cigarette pod nicotine concentration during the 10-puff standardized puff bout and 60-minute ad libitum session.
  After a washout period of at least 48 hours, at lab visit 2 participants receive 1.8% electronic cigarette pod nicotine concentration during the 10-puff standardized puff bout and 60-minute ad libitum session.
  Interventions: Device: Electronic Cigarette with 5% Nicotine Concentration; Device: Electronic Cigarette with 1.8% Nicotine Concentration
- 1.8% Nicotine E-cigarette Followed by 5% Nicotine E-cigarette (Experimental): At lab visit 1 participants receive 1.8% electronic cigarette pod nicotine concentration during the 10-puff standardized puff bout and 60-minute ad libitum session.
  After a washout period of at least 48 hours, at lab visit 2 participants receive 5% electronic cigarette pod nicotine concentration during the 10-puff standardized puff bout and 60-minute ad libitum session.
  Interventions: Device: Electronic Cigarette with 5% Nicotine Concentration; Device: Electronic Cigarette with 1.8% Nicotine Concentration

INTERVENTIONS:
Device: Electronic Cigarette with 5% Nicotine Concentration — Electronic cigarette in 5% nicotine concentration (Vuse Alto), provided for free.
Device: Electronic Cigarette with 1.8% Nicotine Concentration — Electronic cigarette in 1.8% nicotine concentration (Vuse Alto), provided for free.

SUMMARY:
The study will be the first to assess the impact of nicotine concentration on compensatory puffing (total inhaled volume), nicotine delivery, and switch patterns (percent exclusive EC, dual cig-EC, and cig only users) with an explicit focus on AA and White smokers.

DETAILED DESCRIPTION:
1. E-cigarettes (ECs) are projected to exceed combustible cigarette use within two years. Policy makers, health officials, and regulators are concerned that newer nicotine salt-based Ecs that use high concentrations of nicotine in their e-liquids are a major reason for this rapid growth in use. The US Food and Drug Administration (FDA) has regulatory authority to set appropriate tobacco product standards to protect public health and has shown interest in exploring a product standard limiting the level of nicotine in e-liquids. While this regulatory consideration has merit, emerging research suggests it may be misguided, leading to a product that is just as addictive but more harmful. Specifically, among users of earlier, freebase nicotine Ecs (i.e., cig-a-like, tank systems), use of low nicotine e-liquids was associated with a 9-fold increase in e-liquid consumption and all of its related toxicants, likely due to compensatory puffing. The consequences of consuming more e-liquid because of lower nicotine concentration remains an important knowledge gap. Moreover, the National Academies of Science, Engineering, and Medicine have concluded that completely substituting Ecs for cigarettes results in less short-term harm than continued smoking, but the impact of low versus high nicotine concentration e-liquids on a smokers' ability to completely switch to Ecs (versus become 'dual users' or continue smoking) is currently unknown. African American (AA) smokers, who take larger puffs, inhale more intensely, and extract more nicotine and harmful constituents per cigarette smoked, may be particularly impacted by nicotine product standards placed on EC - i.e., greater compensatory puffing and more e-liquid and related toxicant consumption at lower e-liquid concentrations. Unfortunately, the vast majority of information on Ecs and potential product standards come from white populations and have largely ignored African American (AA) smokers who bear a disproportionate burden of tobacco-related morbidity and mortality. As the FDA considers regulatory action to limit the level of nicotine in e-liquids to protect public health, it is critical that research considers vulnerable populations and does not widen disparities.

The long-term goal is to inform a tobacco landscape that will minimize tobacco-related harms and downstream health inequities. The overall objective of this application is to understand the impact of e-liquid nicotine concentration on compensatory puffing, EC and cigarette use patterns (exclusive EC, dual EC-cig, exclusive cig), and resultant exposure to biomarkers of harm among AA and white smokers. Adult AA and white smokers will complete two study phases. In Phase 1, using a randomized crossover design, participants will complete two standardized, 10-puff vaping bouts over 5 mins followed by a 60-minute ad libitum vaping session, using two e-liquids that differ only by nicotine concentration (5% vs. 1.8%) to examine the effect of nicotine concentration on in-lab compensatory puffing, nicotine exposure, and e-liquid consumption. In Phase 2, the same participants will be randomized to 5% or 1.8% nicotine e-liquid and instructed to switch completely for 6 weeks to examine the impact of nicotine concentration on short-term and real-world EC use patterns. The central hypothesis is that, compared to the high nicotine concentration, while vaping the low nicotine concentration, users will engage in compensatory puffing, resulting in greater e-liquid consumption (Phase 1). Moreover, rates of dual use and continued smoking will be higher for the low (versus high) nicotine concentration.

ELIGIBILITY:
Inclusion Criteria:

1. identify as non-Hispanic white or non-Hispanic African American/Black
2. willing to switch from smoking to e-cigarettes for 6 weeks
3. speak and understand English
4. smoke greater than or equal to 25 of the last 30 days for the past 3 months
5. not previously used an e-cigarette for longer than 30 days
6. exhaled carbon monoxide of greater than or equal to 6ppm at screener visit
7. willing to abstain from marijuana for 12 hours prior to in-person lab visits
8. willing to abstain from smoking and vaping for 12 hours prior to 3 in-person lab visits

Exclusion Criteria:

1. weekly use of an EC over the last six months
2. use of tobacco products other than cigarettes on greater than or equal to 10 days in the past 30 days
3. use of EC on more than 5 of the past 30 days
4. current use of cessation medications
5. pregnant, planning to become pregnant, or breastfeeding
6. past 30 day hospitalization/ER visit for psychiatric issue, seizure, stroke, or new heart problem
7. recent history of cardiovascular or pulmonary events in the past three months
8. treatment for alcohol or drug dependence in the past year
9. household member currently or previously enrolled in the study
10. current enrollment in a program aimed at changing smoking patterns

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Leavens, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leavens EL, Driskill LM, Molina N, Eissenberg T, Shihadeh A, Brett EI, Floyd E, Wagener TL. Comparison of a preferred versus non-preferred waterpipe tobacco flavour: subjective experience, smoking behaviour and toxicant exposure. Tob Control. 2018 May;27(3):319-324. doi: 10.1136/tobaccocontrol-2016-053344. Epub 2017 Apr 5. PMID 28381414
- [Background] Wagener TL, Leavens ELS, Mehta T, Hale J, Shihadeh A, Eissenberg T, Halquist M, Brinkman MC, Johnson AL, Floyd EL, Ding K, El Hage R, Salman R. Impact of flavors and humectants on waterpipe tobacco smoking topography, subjective effects, toxicant exposure and intentions for continued use. Tob Control. 2020 May 13:tobaccocontrol-2019-055509. doi: 10.1136/tobaccocontrol-2019-055509. Online ahead of print. PMID 32404518
- [Background] Leavens ELS, Morgan TL, Brett EI, Patzkowsky K, Son J, Molina N, Eissenberg T, Shihadeh A, Leffingwell TR, Wagener TL. Concurrent Alcohol Use and Waterpipe Tobacco Smoking: Smoking Topography, Toxicant Exposure, and Abuse Liability. Nicotine Tob Res. 2020 Feb 6;22(2):280-287. doi: 10.1093/ntr/ntz032. PMID 30820567
- [Background] Leavens ELS, Smith TT, Natale N, Carpenter MJ. Electronic cigarette dependence and demand among pod mod users as a function of smoking status. Psychol Addict Behav. 2020 Nov;34(7):804-810. doi: 10.1037/adb0000583. Epub 2020 Apr 16. PMID 32297753
- [Background] Leavens ELS, Stevens EM, Brett EI, Hebert ET, Villanti AC, Pearson JL, Wagener TL. JUUL electronic cigarette use patterns, other tobacco product use, and reasons for use among ever users: Results from a convenience sample. Addict Behav. 2019 Aug;95:178-183. doi: 10.1016/j.addbeh.2019.02.011. Epub 2019 Feb 18. PMID 30933713
- [Background] Leavens ELS, Stevens EM, Brett EI, Leffingwell TR, Wagener TL. JUUL in school: JUUL electronic cigarette use patterns, reasons for use, and social normative perceptions among college student ever users. Addict Behav. 2019 Dec;99:106047. doi: 10.1016/j.addbeh.2019.106047. Epub 2019 Jul 9. PMID 31442788
- [Background] Wagener TL, Avery JA, Leavens ELS, Simmons WK. Associated Changes in E-cigarette Puff Duration and Cigarettes Smoked per Day. Nicotine Tob Res. 2021 Mar 19;23(4):760-764. doi: 10.1093/ntr/ntaa211. PMID 33049064
- [Background] Stevens EM, Hebert ET, Tackett AP, Leavens ELS, Wagener TL. Harm Perceptions of the JUUL E-Cigarette in a Sample of Ever Users. Int J Environ Res Public Health. 2020 Jul 2;17(13):4755. doi: 10.3390/ijerph17134755. PMID 32630647
- [Background] Wedel AV, Stevens EM, Molina N, Leavens ELS, Roberts C, Wagener TL. Examining pregnant smokers' attitudes toward cessation aids and electronic nicotine delivery systems. J Okla State Med Assoc. 2018 Oct;111(8):812-816. PMID 31404418
- [Background] Waseh S, Dicker AP. Telemedicine Training in Undergraduate Medical Education: Mixed-Methods Review. JMIR Med Educ. 2019 Apr 8;5(1):e12515. doi: 10.2196/12515. PMID 30958269
- [Background] Leavens ELS, Lechner WV, Stevens EM, Miller MB, Meier E, Brett EI, Moisiuc A, Hale JJ, Wagener TL. Electronic cigarette and combustible cigarette use following a campus-wide ban: Prevalence of use and harm perceptions. J Am Coll Health. 2020 May-Jun;68(4):332-335. doi: 10.1080/07448481.2018.1551803. Epub 2019 Jan 25. PMID 30681933
- [Background] Leavens ELS, Meier E, Brett EI, Stevens EM, Tackett AP, Villanti AC, Wagener TL. Polytobacco use and risk perceptions among young adults: The potential role of habituation to risk. Addict Behav. 2019 Mar;90:278-284. doi: 10.1016/j.addbeh.2018.11.003. Epub 2018 Nov 8. PMID 30472536
- [Background] Tackett AP, Leavens ELS, Wiedenmann A, Perez MN, Baker A, Mayes S, Mullins LL, Wagener TL. Preliminary exploration of secondhand smoke exposure in youth with Sickle Cell Disease: biochemical verification, pulmonary functioning, and health care utilization. Psychol Health Med. 2019 Jan;24(1):35-42. doi: 10.1080/13548506.2018.1516294. Epub 2018 Sep 11. PMID 30203658
- [Background] Leavens ELS, Brett EI, Morgan TL, Lopez SV, Shaikh RA, Leffingwell TR, Wagener TL. Descriptive and injunctive norms of waterpipe smoking among college students. Addict Behav. 2018 Feb;77:59-62. doi: 10.1016/j.addbeh.2017.09.006. Epub 2017 Sep 18. PMID 28963891
- [Background] Leavens ELS, Meier E, Tackett AP, Miller MB, Tahirkheli NN, Brett EI, Carroll DM, Driskill LM, Anderson MP, Wagener TL. The impact of a brief cessation induction intervention for waterpipe tobacco smoking: A pilot randomized clinical trial. Addict Behav. 2018 Mar;78:94-100. doi: 10.1016/j.addbeh.2017.10.023. Epub 2017 Oct 28. PMID 29128712
- [Background] Leavens EL, Brett EI, Frank S, Shaikh RA, Leffingwell TR, Croff JM, Wagener TL. Association between breath alcohol concentration and waterpipe lounge patrons' carbon monoxide exposure: A field investigation. Drug Alcohol Depend. 2017 Jan 1;170:152-155. doi: 10.1016/j.drugalcdep.2016.11.010. Epub 2016 Nov 16. PMID 27918950
- [Background] Busch AM, Leavens EL, Wagener TL, Buckley ML, Tooley EM. Prevalence, Reasons for Use, and Risk Perception of Electronic Cigarettes Among Post-Acute Coronary Syndrome Smokers. J Cardiopulm Rehabil Prev. 2016 Sep-Oct;36(5):352-7. doi: 10.1097/HCR.0000000000000179. PMID 27120039
- [Background] Brett EI, Miller MB, Leavens ELS, Lopez SV, Wagener TL, Leffingwell TR. Electronic cigarette use and sleep health in young adults. J Sleep Res. 2020 Jun;29(3):e12902. doi: 10.1111/jsr.12902. Epub 2019 Sep 4. PMID 31486154

RESULTS

PARTICIPANT FLOW:
Groups:
- 5% Nicotine E-cigarette Followed by 1.8% Nicotine E-cigarette: Participants receive a 5% nicotine e-cigarette to use during the 1st vaping session. Following a minimum 48-hour washout period, participants receive a 1.8% nicotine e-cigarette to use during the 2nd vaping session.
- 1.8% Nicotine E-cigarette Followed by 5% Nicotine E-cigarette: Participants receive a 1.8% nicotine e-cigarette to use during the 1st vaping session. Following a minimum 48-hour washout period, participants receive a 5% nicotine e-cigarette to use during the 2nd vaping session.
- Phase 2: 5% Nicotine E-cigarette: Participants randomized to switch to the 5% nicotine e-cigarette in the RCT portion of the study.
- Phase 2: 1.8% Nicotine E-cigarette: Participants randomized to switch to the 1.8% nicotine e-cigarette in the RCT portion of the study.
Period: First Intervention (1 Day)
Arm/Group | 5% Nicotine E-cigarette Followed by 1.8% Nicotine E-cigarette | 1.8% Nicotine E-cigarette Followed by 5% Nicotine E-cigarette | Phase 2: 5% Nicotine E-cigarette | Phase 2: 1.8% Nicotine E-cigarette
Started | 23 | 29 | 0 | 0
Completed | 23 | 29 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Washout (48 Hours)
Arm/Group | 5% Nicotine E-cigarette Followed by 1.8% Nicotine E-cigarette | 1.8% Nicotine E-cigarette Followed by 5% Nicotine E-cigarette | Phase 2: 5% Nicotine E-cigarette | Phase 2: 1.8% Nicotine E-cigarette
Started | 23 | 29 | 0 | 0
Completed | 23 | 25 | 0 | 0
Not Completed | 0 | 4 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | 5% Nicotine E-cigarette Followed by 1.8% Nicotine E-cigarette | 1.8% Nicotine E-cigarette Followed by 5% Nicotine E-cigarette | Phase 2: 5% Nicotine E-cigarette | Phase 2: 1.8% Nicotine E-cigarette
Started | 23 | 25 | 0 | 0
Completed | 23 | 25 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | 5% Nicotine E-cigarette Followed by 1.8% Nicotine E-cigarette | 1.8% Nicotine E-cigarette Followed by 5% Nicotine E-cigarette | Phase 2: 5% Nicotine E-cigarette | Phase 2: 1.8% Nicotine E-cigarette
Started | 23 | 25 | 0 | 0
Completed | 22 | 23 | 0 | 0
Not Completed | 1 | 2 | 0 | 0
Period: Randomized Trial (6 Weeks; 5% vs. 1.8%)
Arm/Group | 5% Nicotine E-cigarette Followed by 1.8% Nicotine E-cigarette | 1.8% Nicotine E-cigarette Followed by 5% Nicotine E-cigarette | Phase 2: 5% Nicotine E-cigarette | Phase 2: 1.8% Nicotine E-cigarette
Started | 0 (Participants were rerandomized at the start of the randomized trial.) | 0 (Participants were rerandomized at the start of the randomized trial.) | 25 | 20
Completed | 0 | 0 | 24 | 19
Not Completed | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- 5% Nicotine E-cigarette Followed by 1.8% Nicotine E-cigarette: At lab visit 1, participants receive a 5% nicotine e-cigarette to use during the vaping session. The researcher and participant were blinded to nicotine concentration during the visit. Following at least a 48-hour washout period, at lab visit 2, participant receive the 1.8% pod for the lab-based vaping session. The researcher and participant were blinded to nicotine concentration during the visit.
- 1.8% Nicotine E-cigarette Followed by 5% Nicotine E-cigarette: At lab visit 1, participants receive a 1.8% nicotine e-cigarette to use during the vaping session. The researcher and participant were blinded to nicotine concentration during the visit. Following at least a 48-hour washout period, at lab visit 2, participant receive the 5% pod for the lab-based vaping session. The researcher and participant were blinded to nicotine concentration during the visit.
- Total: Total of all reporting groups
Arm/Group | 5% Nicotine E-cigarette Followed by 1.8% Nicotine E-cigarette | 1.8% Nicotine E-cigarette Followed by 5% Nicotine E-cigarette | Total
Number analyzed (Participants) | 23 | 29 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (11.9) | 55.9 (9.6) | 55.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 8 | 11 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 15 | 27
  White | 11 | 14 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Inhaled Volume
Description: Differences within participants in total inhaled volume in electronic cigarette puff topography during the pharmacokinetic portions of lab visit 1 and 2
Time Frame: 5 minutes
Population: Data are reported for all participants that completed both lab visits. The number of participants analyzed differs from the number of participants who completed each period/treatment due to missingness of this specific outcome due to equipment malfunction. Data are missing at random and missingness is not systematic.
Measure: Mean (Standard Deviation); unit: mL
Groups:
- 5% Nicotine E-cigarette: Across two lab visits, participants received a 5% nicotine e-cigarette to use during the vaping session. The researcher and participant were blinded to nicotine concentration during the visit.
- 1.8% Nicotine E-cigarette: Across two lab visits, participants received a 1.8% nicotine e-cigarette to use during the vaping session. The researcher and participant were blinded to nicotine concentration during the visit.
Arm/Group | 5% Nicotine E-cigarette | 1.8% Nicotine E-cigarette
Number analyzed (Participants) | 39 | 38
mL | 416.5 (258.3) | 490.3 (255.1)

2. Secondary Outcome: Participant Switch Trajectory
Description: Switch trajectory: biochemically confirmed [exhaled carbon monoxide] complete switch, use of both e-cigarettes and cigarettes, use of only cigarettes, complete cessation [non-use of e-cigarettes and cigarettes with biochemical confirmation]
Time Frame: Week 6 of the Phase 2 period, approximately 8 weeks post-baseline
Measure: Count of Participants; unit: Participants
Groups:
- 5% Nicotine E-cigarette: During randomized trial (phase 2), participants received a 5% nicotine e-cigarette.
- 1.8% Nicotine E-cigarette: During randomized trial (phase 2), participants received a 1.8% nicotine e-cigarette.
Arm/Group | 5% Nicotine E-cigarette | 1.8% Nicotine E-cigarette
Number analyzed (Participants) | 24 | 19
Participants
  complete switch | 10 | 6
  use of both e-cigarettes and cigarettes | 10 | 13
  use of only cigarettes | 3 | 0
  complete cessation | 1 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Safety Population included all participants who received an intervention (i.e., e-cigarette). Total number determined at risk for adverse events is 52.
Groups:
- 5% Nicotine E-cigarette: Participants randomized to switch to 5% e-cigarette.
- 1.8% Nicotine E-cigarette: Participants randomized to switch to 1.8% e-cigarette.
Arm/Group | 5% Nicotine E-cigarette | 1.8% Nicotine E-cigarette
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT05887947/Prot_SAP_000.pdf